CLINICAL TRIAL: NCT07040852
Title: Development and Evaluation of a Mental Health Literacy Intervention in People With Chronic Pain
Brief Title: Learn to Act - Promoting Mental Health Literacy in Chronic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Bárbara Lyrio Ursine, PhD Candidate in Psychology, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.02028.BD
Record Dates: First submitted 2025-06-16; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Mental Health; Health Literacy
Keywords: Chronic Pain; Mental Health Literacy; Health Literacy; Mental Health; pain education
MeSH Terms: conditions — Chronic Pain; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mental Health Literacy Promotion Intervention Program (Experimental): The Intervention Program promoting Mental Health Literacy in people with Chronic Pain is based on the state of the art of Educational Interventions and Mental Health promotion Interventions.
  Interventions: Behavioral: Mental Health Literacy Promotion Intervention Program
- Waitlist Control (Other): Receives intervention later, after initial data collection.
  Interventions: Behavioral: Mental Health Literacy Promotion Intervention Program

INTERVENTIONS:
Behavioral: Mental Health Literacy Promotion Intervention Program — 10 sessions, 90 minutes each, weekly. A face-to-face group treatment for Chronic Pain that focuses on enhancing individuals' understanding of mental health issues, promoting help-seeking behaviors, and reducing stigma associated with mental illness. Intervention includes group discussions, audio-visual material and written material.

SUMMARY:
This pilot randomised controlled trial aims to assess the feasibility, acceptability, and preliminary efficacy of an intervention program promoting Mental Health Literacy. A 10-week group treatment, 90 minutes each session, for adults and older adults with Chronic Pain. Half of the participants will receive the intervention immediately (experimental group), while the other half will not receive it initially. Still, they will receive it after the main phase of the study is completed (control group in waiting list). The intervention focuses on increasing Mental Health Literacy and reducing maladaptive beliefs and behaviours associated with pain. It also explores mechanisms and moderators of change.

DETAILED DESCRIPTION:
Chronic pain is a public health problem that negatively affects well-being and quality of life. In addition to its physiological aspect, pain is a subjective, complex and multidimensional experience. Depression, anxiety, and distress are among the most potent and robust predictors of the transition from acute to chronic pain. Furthermore, maladaptive psychological processes are risk factors for and/or worsening of chronicity and/or intensification of pain symptoms. Therefore, intervention in chronic pain should be a multimodal approach.

Although psychological interventions, particularly Cognitive Behavioral Therapy, are moderately effective in the treatment of pain, the psychoeducational component integrated into these programs has been limited to the biopsychosocial nature of chronic pain and the relationship between psychological distress and pain symptoms, neglecting the promotion of well-being and flourishing. In fact, chronic pain interventions have been almost exclusively limited to reducing symptoms of pain and mental illness, and less so to promoting well-being and overall mental health.

Mental health literacy interventions significantly influence help-seeking behaviours. These interventions, particularly in school settings, show promise in reducing stigma and improving knowledge and attitudes related to mental health. Their efficacy can vary, and there is a need for more tailored approaches to meet the specific needs of individual people. Although Mental Health Literacy is receiving increasing attention as an emerging area of study, it has been an unexplored area in the context of chronic pain. The current study aims to determine the feasibility and evaluate the "Learn to Act" programme -a group-based, mental health literacy intervention in people with chronic pain.

This pilot study seeks to address the following specific research questions: To what extent can the study effectively recruit participants who meet the inclusion criteria? How feasible are the data collection procedures and outcome measures for reaching the target population and evaluating the study objectives? Are the intervention and study procedures acceptable to participants and appropriate for the intended context? Does the research team possess the necessary resources and operational capacity to manage and deliver the intervention effectively? Finally, is the intervention preliminarily effective in increasing mental health literacy, positive affect, satisfaction with life, and quality of life related to spirituality, religiousness and personal beliefs, while reducing pain catastrophising, pain intensity, pain interference, and negative affect? General study design - Participants previously diagnosed with Chronic Pain by a physician will be assigned to two different groups: an experimental group that receives the intervention immediately, and a control group that does not receive the intervention initially but will receive it after the main phase of the study is completed. The feasibility and preliminary efficacy of the Mental Health Literacy Promotion Intervention Program will be assessed by comparing the groups.

Sample: The study will recruit adults and older adults with Chronic Pain. Patients will be provided a study description, a consent form and the research team contact for further clarifications.

The Mental Health Literacy Promotion Intervention Program has the following goals: (a) improve understanding of the pain-mental health connection, (b) reduce mental health stigma, (c) recognize symptoms of mental health challenges, and (d) encourage help-seeking behaviours.

Primary outcomes include changes in Mental Health Literacy and pain catastrophising. Secondary outcomes include quality of life, well-being, satisfaction with life, and pain interference/intensity. The study will assess feasibility through recruitment and retention rates, session attendance, and participant feedback. Mediators and moderators such as pain beliefs, religious coping, meaning in life, and demographic or clinical factors will also be explored to understand the process of change and differential responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 to 64 years old) and seniors (65 years old or older) residing in Portugal.
* Previous diagnosis of Chronic Pain carried out by a doctor.
* Availability to attend sessions.

Exclusion Criteria:

* Active neoplasia.
* Inability to give informed consent (e.g. due to dementia).
* Currently receiving psychological support regularly (sessions > once per semester).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
change from Mental Health Literacy Scale | baseline, immediately post-intervention, and 3-month follow-up
  Mental Health Literacy - higher scores mean more Mental Health Literacy. Minimum value: 35 Maximum value: 160
change from Pain Catastrophizing Scale | baseline, immediately post-intervention, and 3-month follow-up
  Pain Catastrophizing - higher scores mean more catastrophizing thoughts are present.
  Minimum value: 0 Maximum value: 52
change from Brief Pain Inventory - intensity and interference | baseline, immediately post-intervention, and 3-month follow-up
  Pain intensity and interference - higher scores mean more perceived pain severity and interference.
  Minimum value: 0 Maximum value: 10

SECONDARY OUTCOMES:
change from World Health Organization Quality of Life - Spirituality, Religiousness and Personal Beliefs - Bref | baseline, immediately post-intervention, and 3-month follow-up
  Quality of Life Spiritual, Religious and Personal Beliefs - higher scores mean a more positive perception of quality of life in the dimensions of spirituality, religiosity and personal beliefs.
  Minimum value: 9 Maximum value: 45
change from Positive and Negative Affect Schedule | baseline, immediately post-intervention, and 3-month follow-up
  Positive and Negative Affect - higher scores mean more attribution of positive or negative Affect, respectively.
  Minimum value (per subscale): 10 Maximum value (per subscale): 50
change from Satisfaction With Life Scale | baseline, immediately post-intervention, and 3-month follow-up
  Satisfaction With Life - higher scores mean more Satisfaction With Life. Minimum value: 5 Maximum value: 35
change from Brief Religious and Spiritual Coping Scale | baseline, immediately post-intervention, and 3-month follow-up
  Religious and spiritual coping strategies in response to stress and illness.
  * Positive Religious Coping Score (7-28): Higher scores indicate greater reliance on adaptive spiritual coping.
  * Negative Religious Coping Score (7-21): Higher scores reflect significant spiritual struggle and maladaptive coping.
change from Meaning in Life Questionnaire | baseline, immediately post-intervention, and 3-month follow-up
  Presence of Meaning and Search for Meaning - higher scores indicate greater attribution of Presence of Meaning or Search for Meaning, respectively.
  Minimum value (per subscale): 1 Maximum value (per subscale): 25
change from Pain Beliefs and Perceptions Inventory | baseline, immediately post-intervention, and 3-month follow-up
  Pain Beliefs and Perceptions - higher scores mean more attribution of organic or psychological causes of pain.
  Minimum value: 15 Maximum value: 90
Demographics Checklist | baseline
  Gender, age, education level, spirituality/religiousness will be assessed as potential moderators of the intervention's efficacy. These factors may help identify subgroups that respond differently to the intervention.
Clinical Health Profile Checklist | baseline
  Professional healthcare follow-up, comorbid conditions, and pain duration will be assessed as potential moderators of the intervention's efficacy. These factors may help identify subgroups that respond differently to the intervention.
Neuropathic Pain Diagnostic Questionnaire | baseline
  Neuropathic Pain - higher scores mean greater likelihood of neuropathic pain. Minimum value: 0 Maximum value: 7
Cognitive Failures Questionnaire | baseline
  Cognitive Failures - higher scores mean more Cognitive Failures. Minimum value: 0 Maximum value: 100
Patient Global Impression of Change | immediately post-intervention and 3-month follow-up
  Patient's overall perception of change in their health status - higher scores mean the patient's perception that there has been a substantial improvement in their health.
  Minimum value: 1 Maximum value: 7

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Unit/ Anesthesiology Service/ Coimbra Local Health Unit, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No